CLINICAL TRIAL: NCT05208957
Title: Cardiovascular Outcomes and Mortality in Vascular Surgical Patients. A Registry-based Study of in Hospital Mortality and Postoperative Complications in Elective Vascular Surgery at Groote Schuur Hospital
Brief Title: Cardiovascular Outcomes and Mortality in Vascular Surgical Patients
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Christella Alphonsus, Study Principal investigator, University of Cape Town
Other Study IDs: HREC760/2021
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Perioperative Complication; Cardiovascular Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a registry-based study of elective vascular surgical patients undergoing intermediate or high-risk vascular surgical interventions at Groote Schuur hospital, a tertiary academic center, over a 12 month period.

ELIGIBILITY:
Inclusion Criteria:

-

All patients undergoing vascular surgery:

1. 18 years and older
2. Elective procedures
3. Moderate- to high-risk surgical interventions

Exclusion Criteria:

1. Emergency vascular procedures
2. Low risk vascular surgery, i.e. venous stripping
3. All non-vascular surgical interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises all patients, 18 years and older, undergoing any elective moderate- to high-risk vascular surgical intervention at Groote Schuur Hospital. Surgical risk as defined by ESC/ESA 2014 guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Determine in-hospital mortality in elective vascular surgical patients | 12 months

SECONDARY OUTCOMES:
Determine incidence of MACE in elective vascular surgical patients. | 12 months
Describe the risk factors associated with MACE in elective vascular surgical patients | 12 months
Determine incidence of post-operative complications in elective vascular surgical patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christella Alphonsus, MBChB, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared by PI
Supporting Information: Study Protocol, SAP
Time Frame: Not limited
Access Criteria: Contact PI